CLINICAL TRIAL: NCT03616626
Title: Phase III Randomized Study of Adjuvant Whole Breast Versus Partial Breast Irradiation Using Once Daily or Twice Daily Fractionation Scheme in Women With Stage I or II Breast Cancer
Brief Title: Whole Breast Irradiation vs Twice Daily vs. Once Daily Accelerated Partial Breast Irradiation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Rimoun Ramsis Anis Boutrus, Lecturer of Radiation Oncology, National Cancer Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NCI-BC-12/2012
Record Dates: First submitted 2018-07-28; First posted 2018-08-06 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Breast Cancer; Radiation Toxicity
Keywords: Breast Cancer; Accelerated partial Breast Irradiation; Breast cosmesis; radiation Toxicity
MeSH Terms: conditions — Breast Neoplasms; Radiation Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Whole Breast Irradiation (Active Comparator): Adjuvant 3D Conformal Radiation Therapy to a dose of 50 Gy in 25 fractions over 5 weeks. Boost is given as 10 Gy in 5 fractions over one week to patients with high grade tumors or age younger than 50 years
  Interventions: Radiation: Whole Breast Irradiation
- Once Daily APBI (Experimental): Adjuvant 3D Conformal Accelerated Partial Breast Irradiation to a dose of 38.5 Gy in 10 once daily fractions given over 2 weeks
  Interventions: Radiation: Once Daily APBI
- Twice Daily APBI (Experimental): Adjuvant 3D Conformal Accelerated Partial Breast Irradiation to a dose of 38.5 Gy in 10 twice daily fractions given over 1 week
  Interventions: Radiation: Twice Daily APBI

INTERVENTIONS:
Radiation: Once Daily APBI — Adjuvant 3D Conformal Accelerated Partial Breast Irradiation to a dose of 38.5 Gy in 10 once daily fractions given over 2 weeks
  Arms: Once Daily APBI
Radiation: Twice Daily APBI — Adjuvant 3D Conformal Accelerated Partial Breast Irradiation to a dose of 38.5 Gy in 10 twice daily fractions given over 1 week
  Arms: Twice Daily APBI
Radiation: Whole Breast Irradiation — Adjuvant 3D Conformal Radiation Therapy to a dose of 50 Gy in 25 fractions over 5 weeks. Boost is given as 10 Gy in 5 fractions over one week to patients with high grade tumors or age younger than 50 years
  Arms: Whole Breast Irradiation

SUMMARY:
This is a randomized phase III trial in women with invasive carcinoma of the breast with negative axillary nodes treated by Breast Conserving Surgery (BCS). Eligible, patients will be randomly allocated to receive radiotherapy of 3 Dimensional Conformal Radiation Therapy (3DCRT) Whole Breast Irradiation (WBI) 50 Gray (Gy) in 25 daily fractions over 5 weeks or Accelerated Partial Breast Irradiation (APBI) 38.5 Gy in 10 daily fractions of 3.85Gy over two weeks or 38.5 Gy in 10 twice daily fractions of 3.85Gy over one week. Patients will be followed at 6, 12, 18 and 24 months post randomization. Cosmetic outcome will be measured using photographs and evaluated by a panel of trained radiation oncologists. Radiation toxicity will be assessed using National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE).

DETAILED DESCRIPTION:
Women with invasive carcinoma of the breast less than 3 cm with negative axillary nodes , following BCS, who meet the inclusion criteria will be approached for potential study enrollment.

Eligible, consenting patients will be randomly allocated to receive radiotherapy of 3DCRT WBI 50 Gy in 25 fractions over 5 weeks or APBI 38.5 Gy in 10 once daily fractions of 3.85Gy over two weeks or 38.5 Gy in 10 twice daily fractions of 3.85 Gy over one week. Patients will be followed at 6, 12, 18 and 24 months post randomization. Cosmetic outcome will be measured using photographs and evaluated by a panel of trained radiation oncologists using the EORTC Breast Cosmetic Rating System. Radiation toxicity will be assessed using the NCI CTCAE version 4.0. The primary outcome is to compare the acute, late toxicities and adverse cosmetic outcomes at 6, 12 and 18 months among the three groups.

ELIGIBILITY:
Inclusion Criteria:

Tumor characteristics

* Histologically confirmed invasive adenocarcinoma of the breast
* Tumors must be ≤ 3 cm. Gross disease must be unifocal. Negative lymph nodes
* Hormone receptor status:

Estrogen receptor (ER) status known Progesterone status known if ER analysis is negative Marginal or borderline results are considered positive Surgery

* Tumor removed with conservative breast surgery with adequate margin
* Re-excision of surgical margins allowed
* No prior breast implants
* Prior axillary staging required for patients including 1 of the following:

  * Sentinel node biopsy alone (if sentinel node is negative)
  * Sentinel node biopsy followed by axillary dissection if sentinel node is positive)
  * Axillary dissection alone with ≥ 6 axillary nodes
* Target lumpectomy cavity clearly delineated AND target lumpectomy/whole breast reference volume ≤ 30% based on postoperative pre-randomization CT scan
* Final surgery (i.e., lumpectomy, re-excision of margins, or axillary staging procedure) within the past 42 days
* No prior biologic therapy for this malignancy Chemotherapy
* No prior chemotherapy for this malignancy
* No concurrent chemotherapy during study radiotherapy Endocrine therapy
* No prior hormonal therapy for this malignancy
* Concurrent hormonal therapy allowed provided it is not administered during chemotherapy
* No concurrent raloxifene, tamoxifen, or other selective estrogen receptor modulating drugs
* No concurrent hormone replacement therapy Radiotherapy
* No prior radiotherapy for this malignancy
* No prior breast or thoracic radiotherapy
* No concurrent regional nodal irradiation Other
* No other concurrent anticancer therapy Menopausal status
* Premenopausal or postmenopausal Performance status
* WHO 0-1 Other
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective non-hormonal contraception

Exclusion Criteria:

* Multicentric carcinoma in more than 1 quadrant or separated by ≥ 4 cm.
* Non-epithelial breast malignancies (e.g., sarcoma or lymphoma).
* Positive axillary nodes.
* Palpable or radiographically suspicious ipsilateral or contralateral axillary, supraclavicular, infraclavicular, or internal mammary nodes unless there is histologic confirmation that these nodes are negative for tumor.
* Suspicious microcalcifications, densities, or palpable abnormalities in the ipsilateral or contralateral breast unless biopsied and found to be benign
* Paget's disease of the nipple
* Previous history of invasive breast cancer or DCIS.
* Synchronous bilateral invasive or non-invasive breast cancer
* Collagen vascular disease (e.g., systemic lupus erythematosus or scleroderma), specifically dermatomyositis with a CPK level above normal, or active skin rash
* Psychiatric or addictive disorder that would preclude study therapy

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2013-07-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in the Adverse cosmetic outcome using the EORTC Breast Cosmetic Rating System | prior to radiation, 6,12 and 18 months after radiation
  The primary outcome is the change in the adverse cosmesis assessed prior to radiation, 6, 12 and 18 months after end of radiation. The cosmetic outcome will be assessed by a radiation oncologist who is unaware of treatment allocation, using the EORTC Breast Cosmetic Rating System.

SECONDARY OUTCOMES:
Ipsilateral Breast Tumor Recurrence (IBTR) | throughout the study up to 5 years
  defined as recurrent invasive or in situ cancer in the ipsilateral breast. Histological evidence of local recurrence will be required.
Disease Free Survival | throughout the study up to 5 years
  defined as the time from randomization to the time of documented recurrent disease in the ipsilateral breast or regional nodes (supraclavicular, axillary or internal mammary) or distant sites (e.g. bone, liver, lung or brain).
Overall Survival | From date of randomization until the date of death up to 5 years
  defined as the time from randomization to death from any cause
Radiation Induced Early and late toxicities | during radiation and at 6, 12 and 18 months after radiation
  using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v.4.0

CONTACTS AND LOCATIONS:
Overall Officials: Rimoun Boutrus, M.D., Principal Investigator — Radiation Oncology Department, National Cancer Institute, Cairo University
Locations (1):
- National Cancer Institute, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Hepel JT, Tokita M, MacAusland SG, Evans SB, Hiatt JR, Price LL, DiPetrillo T, Wazer DE. Toxicity of three-dimensional conformal radiotherapy for accelerated partial breast irradiation. Int J Radiat Oncol Biol Phys. 2009 Dec 1;75(5):1290-6. doi: 10.1016/j.ijrobp.2009.01.009. Epub 2009 Apr 22. PMID 19395195
- [Result] Jagsi R, Ben-David MA, Moran JM, Marsh RB, Griffith KA, Hayman JA, Pierce LJ. Unacceptable cosmesis in a protocol investigating intensity-modulated radiotherapy with active breathing control for accelerated partial-breast irradiation. Int J Radiat Oncol Biol Phys. 2010 Jan 1;76(1):71-8. doi: 10.1016/j.ijrobp.2009.01.041. PMID 19409733
- [Result] Vicini F, Winter K, Wong J, Pass H, Rabinovitch R, Chafe S, Arthur D, Petersen I, White J, McCormick B. Initial efficacy results of RTOG 0319: three-dimensional conformal radiation therapy (3D-CRT) confined to the region of the lumpectomy cavity for stage I/ II breast carcinoma. Int J Radiat Oncol Biol Phys. 2010 Jul 15;77(4):1120-7. doi: 10.1016/j.ijrobp.2009.06.067. Epub 2009 Nov 10. PMID 19910132
- [Result] Chen PY, Wallace M, Mitchell C, Grills I, Kestin L, Fowler A, Martinez A, Vicini F. Four-year efficacy, cosmesis, and toxicity using three-dimensional conformal external beam radiation therapy to deliver accelerated partial breast irradiation. Int J Radiat Oncol Biol Phys. 2010 Mar 15;76(4):991-7. doi: 10.1016/j.ijrobp.2009.03.012. Epub 2009 Jun 8. PMID 19515514
- [Result] Goyal S, Daroui P, Khan AJ, Kearney T, Kirstein L, Haffty BG. Three-year outcomes of a once daily fractionation scheme for accelerated partial breast irradiation (APBI) using 3-D conformal radiotherapy (3D-CRT). Cancer Med. 2013 Dec;2(6):964-71. doi: 10.1002/cam4.157. Epub 2013 Oct 31. PMID 24403270
- [Result] DE Paula U, D'Angelillo RM, Barbara R, Caruso C, Gomellini S, Caccavari A, Costarelli L, Scavina P, Mauri M, Santini E, Antonaci A, Cavaliere F, LA Pinta M, Loreti A, Fortunato L. Once Daily Accelerated Partial Breast Irradiation: Preliminary Results with Helical Tomotherapy(R). Anticancer Res. 2016 Jun;36(6):3035-9. PMID 27272823
- [Result] Bentzen SM, Yarnold JR. Reports of unexpected late side effects of accelerated partial breast irradiation--radiobiological considerations. Int J Radiat Oncol Biol Phys. 2010 Jul 15;77(4):969-73. doi: 10.1016/j.ijrobp.2010.01.059. No abstract available. PMID 20610037